CLINICAL TRIAL: NCT02192216
Title: The Effect of Resistance Training and Aerobic Training on Body Composition During Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting issues and limited personel ressources
Sponsor: Department of Public Health, Denmark (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Simon Lønbro, M.Sc., PhD., Department of Public Health, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SKDM2014; 41408 (Other: Denmark: Ethics Committee)
Record Dates: First submitted 2014-07-04; First posted 2014-07-16 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Neoplasms
Keywords: Body composition; Chemotherapy; Muscle mass; Muscle function; Exercise
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise & Chemotherapy (Experimental): Following a control period during active chemotherapy the patients undergo ten weeks of supervised exercise comprised of resistance and aerobic training in combination with protein supplementation during ongoing chemotherapy.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise
  Other Names: Resistance training; Aerobic exercise; Protein supplementation

SUMMARY:
Chemotherapy can induce muscle loss in colorectal, breast and advanced renal cell carcinoma patients. The Danish nation-wide training and rehabilitation offer 'Body & Cancer' offers intensive resistance and endurance training to all Danish cancer patients receiving chemotherapy with the aim of reducing treatment-related fatigue and physical impairments, but the potential of the training to preserve or improve muscle mass is uninvestigated.

Furthermore, the underlying biological mechanisms of treatment and/or exercise induced changes in muscle mass in cancer patients remains uninvestigated.

Thus, the primary purpose of the present study is to investigate changes in body composition during chemotherapy and after resistance and aerobic training combined with protein supplementation during ongoing chemotherapy in cancer patients. Secondly, we aim to investigate the underlying biological mechanisms of muscle mass regulation in biopsies obtained before and after a control period as well as after 10 weeks of exercise, both during chemotherapy.

We hypothesize that 10 weeks exercise will improve muscle mass and body composition in cancer patients during chemotherapy as compared to a control period during chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving curative, adjuvant, neo-adjuvant or palliative chemotherapy
* No documented bone metastases or myelomatosis
* No documented CNS affection
* WHO performance status 0-1
* No chronical thrombocytopenia or leukopenia
* No physical conditions preventing exercise participation
* No serious symptoms of heart disease
* No dementia or mental illness preventing participation
* Signed written concent
* Age above 18 years

Exclusion Criteria:

* Participation in systematic resistance training three months prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes in body composition | Assessment before (baseline) and after (pre-training) the control period of 7 weeks (average), where patients recieve chemotherapy, and again after completion of 10 weeks of exericse (post-training).
  Changes in lean body mass and fat mass wil be assessed using Dual Energy X-Ray Absorptiometry

SECONDARY OUTCOMES:
Changes in underlying biological mechanisms associated with changes in muscle mass | Assessment before (baseline) and after (pre-training) the control period of 7 weeks (average), where patients recieve chemotherapy, and again after completion of 10 weeks of exericse (post-training).
  Analyzed from muscle biopsies from m. vastus lateralis and venous blood samples
Changes in dynamic muscle strength | Assessment before (baseline) and after (pre-training) the control period of 7 weeks (average), where patients recieve chemotherapy, and again after completion of 10 weeks of exericse (post-training).
  Changes in muscle strength will be assessed using 1 repetition maximum (kg) tests using conventional training equipment.
Changes in aerobic performance | Assessment before (baseline) and after (pre-training) the control period of 7 weeks (average), where patients recieve chemotherapy, and again after completion of 10 weeks of exericse (post-training).
  Changes in aerobic performance will be assessed using the Watt max bicycle ergometer test. Maximal oxygen consumption (L O2 pr min) will be estimated based on this test.
Changes in cancer related fatigue and quality of life | Assessment before (baseline) and after (pre-training) the control period of 7 weeks (average), where patients recieve chemotherapy, and again after completion of 10 weeks of exericse (post-training).
  Changes in cancer related fatigue and quality of life wil be assessed using the European Organisation for Research and Treatment of Cancer (EORTC) questionaire QLQ C30
Changes in functional performance | Assessment before (baseline) and after (pre-training) the control period of 7 weeks (average), where patients recieve chemotherapy, and again after completion of 10 weeks of exericse (post-training).
  Changes in functional performance will be assessed using various validated functional performance tests. Thus, changes will be asssessed in 30 s arm curl test (max repetitions) , 30 s chair rise test (max repetitions), stair climbing test (time to ascend to flights of stairs), 10 m maximal gait speed test (time to walk 10 m as fast as possible).

CONTACTS AND LOCATIONS:
Overall Officials: Simon Loenbro, M.Sc., PhD, Principal Investigator — Dept. of Public Health, Sect. for Sports Science, Aarhus University
Locations (1):
- Dept of Oncology, Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- [Derived] Moller AB, Lonbro S, Farup J, Voss TS, Rittig N, Wang J, Hojris I, Mikkelsen UR, Jessen N. Molecular and cellular adaptations to exercise training in skeletal muscle from cancer patients treated with chemotherapy. J Cancer Res Clin Oncol. 2019 Jun;145(6):1449-1460. doi: 10.1007/s00432-019-02911-5. Epub 2019 Apr 9. PMID 30968255